CLINICAL TRIAL: NCT01656343
Title: Belatacept and Risk of PTLD in US Renal Transplant Recipients
Brief Title: Belatacept and Risk of Post-transplant Lymphoproliferative Disorder in US Renal Transplant Recipients
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: IM103-075
Record Dates: First submitted 2012-07-31; First posted 2012-08-03 (Estimated); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Kidney Transplantation; Transplantation, Kidney
MeSH Terms: interventions — Calcineurin Inhibitors; Abatacept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Belatacept treated kidney-only transplant recipients
  Interventions: Drug: Belatacept
- CNI treated kidney-only transplant recipients
  Interventions: Drug: Calcineurin inhibitors (CNI)

INTERVENTIONS:
Drug: Calcineurin inhibitors (CNI) — No Intervention
  Groups: CNI treated kidney-only transplant recipients
Drug: Belatacept — No Intervention
  Other Names: Nulojix
  Groups: Belatacept treated kidney-only transplant recipients

SUMMARY:
* To estimate the incidence rates of post-transplant lymphoproliferative disorder (PTLD) in adult, EBV seropositive, kidney alone transplant recipients treated with belatacept at the time of transplantation
* To estimate the incidence rates of PTLD in adult, EBV seropositive, kidney alone transplant recipients treated with calcineurin inhibitors (CNI)-based regimens at the time of transplantation
* To compare the PTLD incidence rates in adult, EBV seropositive, kidney alone transplant recipients treated with belatacept to the rates in adult, EBV seropositive, kidney alone transplant recipients treated with CNI-based regimens at the time of transplantation

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com.

Inclusion Criteria:

* Adult,
* EBV seropositive, Kidney only transplant recipients initiated on belatacept and adult,
* EBV seropositive, kidney only transplant recipients initiated on CNIs reported to the United Network for Organ Sharing (UNOS) during the period of recruiting belatacept users

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult, EBV seropositive, kidney only transplant recipients initiated on belatacept and adult, EBV seropositive, kidney only transplant recipients initiated on CNIs reported to the UNOS during the period of recruiting belatacept users
Sampling Method: Non-Probability Sample
Enrollment: 775 (Actual)
Dates: Start 2011-10-31 (Actual); Primary Completion 2019-08-05 (Actual); Study Completion 2019-08-05 (Actual)

PRIMARY OUTCOMES:
Incidence rates of post-transplant lymphoproliferative disorder (PTLD) in adult, EBV seropositive, kidney alone transplant recipients treated with belatacept at the time of transplantation | Every 6 months for up to 72 months
Incidence rates of PTLD in adult, EBV seropositive, kidney alone transplant recipients treated with calcineurin inhibitors (CNI)-based regimens at the time of transplantation | Every 6 months for up to 72 months
Ratio for PTLD incidence rates in adult, EBV seropositive, kidney alone, belatacept treated patients and adult EBV seropositive, kidney alone, CNI-treated patients at the time of transplantation | Every 6 months for up to 72 months

SECONDARY OUTCOMES:
Incidence rates of PTLD in subgroups of belatacept-treated, adult, kidney alone transplant recipients defined by recipient Epstein-Barr virus (EBV) serostatus (negative or unknown) and by donor to recipient EBV serostatus | Every 6 months for up to 72 months
Ratio for PTLD incidence rates in the belatacept-treated subgroups defined by EBV serostatus (negative or unknown) to the rates in corresponding CNI-treated subgroups | Every 6 months for up to 72 months
Incidence rates of PTLD in subgroups of belatacept-treated, adult, kidney alone transplant recipients defined by recipient cytomegalovirus (CMV) serostatus and by donor to recipient CMV serostatus | Every 6 months for up to 72 months
Ratio for PTLD incidence rates in the belatacept-treated subgroups defined by CMV serostatus to the rates in corresponding CNI-treated subgroups | Every 6 months for up to 72 months
Characteristics (age, gender, weight, BMI, use of immunosuppressive medications, and type of induction medications) of PTLD cases, and the location and mortality of PTLD | Every 6 months for up to 72 months
  Characteristics in adult, kidney alone transplant recipients treated with belatacept at transplantation and in subgroups of these transplant recipients defined by EBV serostatus and CMV serostatus
Ratio for characteristics of PTLD cases, and the location and mortality of PTLD, in adult, kidney alone transplant recipients treated with belatacept at transplantation to those treated with CNI-based regimens at transplantation | Every 6 months for up to 72 months
Two year incidence rates of PTLD by calendar year of transplantation in adult, kidney alone transplant recipients treated with belatacept at transplantation, and in subgroups of these transplant recipients defined by EBV serostatus and by CMV serostatus | Every 6 months for up to 24 months
Incidence rates of PTLD by immunosuppressive regimen changes in adult, kidney alone transplant recipients who switch to or from belatacept during the period from transplant to the end of one-year follow-up | Every 6 months for up to 12 months follow up

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

REFERENCES:
- [Derived] Cherikh WS, Kou TD, Foutz J, Baker TJ, Gomez-Caminero A. Patterns of belatacept use and risk of post-transplant lymphoproliferative disorder in US kidney transplant recipients: An analysis of the Organ Procurement and Transplantation Network database. PLoS One. 2025 Jan 10;20(1):e0311935. doi: 10.1371/journal.pone.0311935. eCollection 2025. PMID 39792912
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome